CLINICAL TRIAL: NCT04840173
Title: Beyond Listening: A Music-based Caregiver Intervention
Brief Title: Beyond Listening: A Music-based Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: MJHS Institute for Innovation in Palliative Care (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MJHSPalliative
Record Dates: First submitted 2021-04-07; First posted 2021-04-09 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Alzheimer's Disease (Incl Subtypes); Depressive Symptoms
Keywords: Music Therapy; Music Interventions; Caregiver Singing; Family Caregivers; Dementia; Alzheimer's Disease; ADRD; Neuropsychiatric symptoms; Therapeutic music; Non-pharmacological interventions; Creative arts therapy; Vascular dementia; Behavioral and Psychological symptoms of dementia; Caregiver Burden; Depression; Agitation; Mood; Pleasure
MeSH Terms: conditions — Alzheimer Disease; Depression; Dementia; Dementia, Vascular; Behavior; Caregiver Burden; Psychomotor Agitation | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music at home (Experimental): Caregivers will use Singing, music listening, or moving with music twice a week for 30 minutes with their care recipient.
  Interventions: Behavioral: Music

INTERVENTIONS:
Behavioral: Music — During attendance at a one hour, 6-week psychosocial classroom or virtual training, caregivers will learn to use singing and other music-based interventions, implementing them each week before the informational session.

SUMMARY:
Study will be conducted to determine if caregivers who use music at home will feel less burden and whether the person they are caring for will demonstrate decreased symptoms of dementia. Caregivers will participate in a series of psycho-educational trainings for six weeks. During this time, caregivers will learn how to use singing, music listening and music with movement with their family member. Caregivers should feel less stressed and a decreased sense of burden. The care recipient should appear happier with less occurrences of depression or restlessness.

DETAILED DESCRIPTION:
Our study will incorporate caregivers and their care receivers who are diagnosed with dementia and agitation co-occurring depression. The primary study outcomes are the following: caregiver burden, measured with the Zarit Caregiver Burden Intervention; mood, measured with the Cornell-Brown Scale for Quality of Life; agitation, measured with the Neuropsychiatric Inventory Questionnaire; and focus group and diaries will be used to gain a descriptive account of caregiver experiences of facilitation of music intervention. Assessment time frame is focus group with caregivers, then pre-tests for baseline. Before the first workshop, caregivers will be asked to participate in a focus group with other caregivers.

Following pre-tests and focus group, caregivers will participate in a 6-week classroom workshop including the following topics: adding singing and music with movement to address mood or agitation, music listening to assist with transitions or difficult tasks, implementing background music for compliance during activities of daily living, creating individualized playlists/interventions to address undesirable behaviors, and the use of an MP3 player . The 6-week workshop will take place in person or via Zoom. Potential participants will be asked to meet for an hour, once weekly.

During the workshops, caregivers will be taught music-based interventions that involve adding singing and music with movement to address mood or agitation, music listening to assist with transitions or difficult tasks, background music for compliance and the creation of individualized playlists to address undesirable behaviors.

This psychosocial intervention will teach caregivers to incorporate a music-based intervention. The music-based intervention is a non-invasive program that involves singing, music with movement and music listening.

During these 6 weeks, caregivers will implement the music intervention with the care recipient and document weekly diaries. There will be a 3 month follow up designated for participants to repeat the completion of the questionnaires, Zarit Caregiver Burden Interview, Cornell-Brown Scale for Quality of Life, and Neuropsychiatric Inventory Questionnaire. These questions will be about participants' moods, agitation level or caregiver burden. This information will be collected in person at Menorah from potential caregiver participants. Principal Investigator will call to gather this data from the caregivers.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of dementia,
* person with dementia exhibits neuropsychiatric symptoms of dementia such as agitation, restlessness, depressed mood, etc.,
* A family member or close friend of a person with dementia,
* Family member must be able to read or write in basic English.

Exclusion Criteria:

* Diagnosis or history of mental illness
* Inadequate hearing even with corrective device
* History of psychosis or other mental disorders other than depression
* History or presence of substance or alcohol abuse.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Mean of 12-item Zarit Caregiver Burden Interview at Week 6. The minimum score is 0 and maximum score is 88. | Baseline, week 6 and month three
  The Zarit Caregiver Burden is a validated, self-reported instrument assessing personal strain and role strain of family caregiver. Higher scores suggest more caregiver burden.
Change from Baseline Quality of Life on the 19-item Cornell-Brown Scale for Quality of Life at Week 6. . | Baseline, week 6 and month three
  The Cornell-Brown Scale for Quality of Life is a validated measure assessing mood related bi-polar items such as anxiety vs comfort, sadness vs happiness, irritability vs tolerance, etc. for care recipients. This is completed by the caregiver on behalf of the care recipient. The minimum score for this measure is -38 and the maximum score is 38. A higher score indicates higher quality of life.
Change from baseline symptoms on the 12-item Neuropsychiatric Inventory Questionnaire at Week 6. | Baseline, week 6 and month three
  The Neuropsychiatric Inventory Questionnaire is a validated measure completed by the caregiver on behalf of the care recipient assessing neuropsychiatric symptoms and behaviors associated with dementia. The scores range from 0 to 36 for individual symptoms. Higher scores indicate higher degrees of severity. Caregiver distress scores range from 0 to 55 with higher scores indicating higher distress.

SECONDARY OUTCOMES:
Qualitative description of usefulness of music intervention | Diaries will be collected at week 6
  Caregivers will be asked to keep weekly diaries of their use of music with care recipient.

CONTACTS AND LOCATIONS:
Locations (1):
- Menorah Center for Nursing and Rehabilitation, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be shared.
Supporting Information: Study Protocol
Time Frame: The study protocol will be available following the study for one year.
Access Criteria: Individuals interested in accessing the study protocol can reach out to the PI via email at kray@mjhs.org

REFERENCES:
- [Background] Ziv N, Granot A, Hai S, Dassa A, Haimov I. The effect of background stimulative music on behavior in Alzheimer's patients. J Music Ther. 2007 Winter;44(4):329-43. doi: 10.1093/jmt/44.4.329. PMID 17997624
- [Result] Gerdner LA. Individualized music for dementia: Evolution and application of evidence-based protocol. World J Psychiatry. 2012 Apr 22;2(2):26-32. doi: 10.5498/wjp.v2.i2.26. PMID 24175165
- [Result] Kaufer DI, Cummings JL, Ketchel P, Smith V, MacMillan A, Shelley T, Lopez OL, DeKosky ST. Validation of the NPI-Q, a brief clinical form of the Neuropsychiatric Inventory. J Neuropsychiatry Clin Neurosci. 2000 Spring;12(2):233-9. doi: 10.1176/jnp.12.2.233. PMID 11001602
- [Result] Ray KD, Mittelman MS. Music therapy: A nonpharmacological approach to the care of agitation and depressive symptoms for nursing home residents with dementia. Dementia (London). 2017 Aug;16(6):689-710. doi: 10.1177/1471301215613779. Epub 2015 Oct 29. PMID 26519453
- [Result] Ready RE, Ott BR, Grace J, Fernandez I. The Cornell-Brown Scale for Quality of Life in dementia. Alzheimer Dis Assoc Disord. 2002 Apr-Jun;16(2):109-15. doi: 10.1097/00002093-200204000-00008. PMID 12040306
- [Result] Sarkamo T, Tervaniemi M, Laitinen S, Numminen A, Kurki M, Johnson JK, Rantanen P. Cognitive, emotional, and social benefits of regular musical activities in early dementia: randomized controlled study. Gerontologist. 2014 Aug;54(4):634-50. doi: 10.1093/geront/gnt100. Epub 2013 Sep 5. PMID 24009169
- [Result] Zarit SH, Reever KE, Bach-Peterson J. Relatives of the impaired elderly: correlates of feelings of burden. Gerontologist. 1980 Dec;20(6):649-55. doi: 10.1093/geront/20.6.649. No abstract available. PMID 7203086